CLINICAL TRIAL: NCT00762450
Title: Effect on Bacterial Glycolytic Acid Formation on Plaque
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2008-PLA-01-AM
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2011-02-15 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Triclosan; Fluorides; hydrated silica gel-based toothpaste; Amino Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A- Positive Control (Active Comparator): fluoride/triclosan/copolymer toothpaste
  Interventions: Drug: Triclosan, Fluoride
- B - Silica control (Placebo Comparator): fluoride only toothpaste
  Interventions: Drug: fluoride
- C- Experimental product (Experimental): fluoride/triclosan/amino acid toothpaste
  Interventions: Drug: Fluoride, triclosan, amino acid

INTERVENTIONS:
Drug: Triclosan, Fluoride — Rinse 3 times daily with assigned toothpaste slurry
  Other Names: Total+ Whitening toothpaste
  Arms: A- Positive Control
Drug: fluoride — Rinse 3 times daily with assigned toothpaste slurry
  Other Names: placebo toothpaste (No triclosan, no amino acid)
  Arms: B - Silica control
Drug: Fluoride, triclosan, amino acid — Rinse 3 times daily with assigned toothpaste slurry
  Arms: C- Experimental product

SUMMARY:
To determine the effect of an amino acid on bacterial glycolytic acid formation in human interdental plaque.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary dentition is preferentially natural.
* Maxillary restorations and/or reconstructions and eventual partial dentures must be in clinically good condition.
* Natural mandibular front teeth and first premolars (4-4) are retained.
* Second mandibular molars are ideally present to serve as abutment teeth.
* Mandibular restorations and/or reconstructions must be in clinically good condition.
* Partial mandibular denture replacing second premolars and first (and second) molars in good clinical condition.
* Subjects should have a stimulated saliva flow rate of 1-2 ml/min (by chewing paraffin wax).
* Willingness to give their informed consent and comply with the protocol.
* No history of allergy to personal/oral care consumer products or ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study

Exclusion Criteria:

* Current participation in other dental clinical trials.
* Subjects who are unable to provide sufficient plaque growth over a 2-day non- brushing period (by visual assessment).
* Subjects in whom the plaque pH fails to fall sufficiently, i.e. at least to pH 5 following a sucrose rinse.
* Subjects with poor oral health, i.e. with advanced periodontitis, un-restored carious lesions and stomatological diseases.
* Subjects taking drugs known to currently affect salivary flow.
* Subjects with un-stimulated salivary flow <0.3 ml/min and/or stimulated flow <0.9 ml/min.
* Women who are pregnant or breastfeeding
* History of allergy to common dentifrice ingredients
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)
* Women of child bearing potential and not on birth control (Diaphragm, birth control pills or implants, IUD (intrauterine device) or condoms)
* Medical condition which requires premedication prior to dental procedures/visits
* History of allergy to amino acids

Ages: 72 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Imfeld, MBA, Principal Investigator
Locations (1):
- University of Zurich, Dental Institute Dept. of Preventive, Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects are recruited by the PI at the clinical site
Pre-assignment Details: subjects are screened for medical and oral health criteria and start a 1 week washout period.
Groups:
- Placebo 1st, Active Comparator 2nd and Experimental Last; Active Comparator 1st, Experimental 2nd and Placebo Last; Experimental 1st, Placebo 2nd and Active Comparator Last: Order of study treatment toothpastes for the enrolled panelist placed in that treatment group. All panelists brushed their teeth with all study treatments, just the order of appearance changed. All panelists rinsed their mouths with a slurry of the assigned toothpaste three times a day for 7 days.
Period: 1st Treatment Period
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental Last | Active Comparator 1st, Experimental 2nd and Placebo Last | Experimental 1st, Placebo 2nd and Active Comparator Last
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Washout After 1st Treatment Period
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental Last | Active Comparator 1st, Experimental 2nd and Placebo Last | Experimental 1st, Placebo 2nd and Active Comparator Last
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: 2nd Treatment Period
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental Last | Active Comparator 1st, Experimental 2nd and Placebo Last | Experimental 1st, Placebo 2nd and Active Comparator Last
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Washout After 2nd Treatment Period
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental Last | Active Comparator 1st, Experimental 2nd and Placebo Last | Experimental 1st, Placebo 2nd and Active Comparator Last
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: 3rd Treatment Period
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental Last | Active Comparator 1st, Experimental 2nd and Placebo Last | Experimental 1st, Placebo 2nd and Active Comparator Last
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Positive Control Second and Experimental Last | Positive Control First, Experimental Second and Placebo Last | Experimental First, Placebo Second and Positive Control Last | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 2 | 2 | 2 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 76.5 (3.5) | 77.5 (0.7) | 73.5 (2.1) | 75.8 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Switzerland | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: ph of Dental Plaque After Sucrose Challenge
Description: Panelists rinsed with toothpaste slurry (2 grams of toothpaste dissolved in 10 ml of water) waited 20 minutes and then rinsed with a 10% sucrose solution. Sucrose challenge is used to change the ph in the mouth and help determine if the toothpastes used in this study and control dental plaque growth.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: ph of dental plaque
Arm/Group | Active Comparator | Placebo - Silica Control | Experimental Toothpaste
Number analyzed (Participants) | 6 | 6 | 6
ph of dental plaque | 4.88 (0.38) | 5.04 (0.38) | 4.98 (0.24)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo - Silica Control vs Experimental Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA; paired t-tests

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Placebo First, Positive Control Second and Experimental Last | Positive Control First, Experimental Second and Placebo Last | Experimental First, Placebo Second and Positive Control Last
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less